CLINICAL TRIAL: NCT01490320
Title: The Effect of Primary Care Interventions on Children's Media Viewing Habits and Exposure to Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Seth Scholer, Associate Professor of Pediatrics, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB# 100401
Record Dates: First submitted 2011-12-07; First posted 2011-12-12 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Violence
Keywords: Violence prevention; Media; Primary care; Parenting
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Parents in control group experienced a routine primary care visit.
  Interventions: Other: Control Group
- Handout intervention (Experimental): Caregivers assigned to the hand-out group were instructed to read the AAP hand-out "Pulling the Plug On TV Violence." This 2 page hand-out emphasizes the negative effect that television has on children's behavior and makes recommendations about limiting media. The RA did not supervise the reading of the handout.
  Interventions: Behavioral: AAP Handout entitled, Pulling the Plug on Violence.
- Multimedia intervention (Experimental): Caregivers assigned to the multimedia group were instructed to watch "Recommendation 3: Decrease Exposure to Violence" from the Play Nicely program, a 5 minute video in English and Spanish that teaches caregivers about the negative impact of violent media and instructs parents about the importance of limiting media. The intervention was presented to the parents on a mobile laptop computer.
  Interventions: Behavioral: Play Nicely Program

INTERVENTIONS:
Behavioral: AAP Handout entitled, Pulling the Plug on Violence. — This handout is two pages and is part of the Connected Kids Program, American Academy of Pediatrics
  Arms: Handout intervention
Behavioral: Play Nicely Program — Multimedia program available at www.playnicely.org.
  Arms: Multimedia intervention
Other: Control Group — Standard care in primary care clinic.
  Arms: Control

SUMMARY:
The American Academy of Pediatrics recommends that parents receive anticipatory guidance about violence prevention as part of the routine well child visit. Educational resources are needed to help physicians routinely provide these important anticipatory guidance messages. In this study, consecutive parents will be exposed to routine anticipatory guidance messages before the well child visit with the physician. After the clinic visit, parents will be invited to participate in a research study to determine if they plan any changes at home. The key research question of this study is:

Can a brief multimedia program (i.e. Play Nicely program) and/or the AAP Connected Kids brochure, entitled, "Pulling the Plug on TV Violence", help parents develop plans to decreases their children's exposure to violence in the media (e.g. less media time, no TV in the bedroom)?

ELIGIBILITY:
Inclusion Criteria:

* Participants included English and Spanish speaking caregivers of 2-12 year old children presenting to the pediatric primary care clinic for a well-child visit.

Exclusion Criteria:

* Parents who could not speak either English or Spanish.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Changes in media viewing habits | Baseline and 2-4 weeks
  At the 2 week follow up phone call, parents were asked:
  "Since your clinic visit, have you made any changes related to your child's media viewing habits such as TV, movies, or computer games?"
Changes in exposure to violence. | Baseline and 2-4 weeks
  At the 2 week follow up phone call, parents were asked:
  "Since your clinic visit, have you made any changes related to decreasing your child's exposure to violence, either violence in the media or violence at home?"

CONTACTS AND LOCATIONS:
Overall Officials: Seth J Scholer, MD, MPH, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Pediatric Primary Care Clinic, Nashville, Tennessee, United States

REFERENCES:
- [Background] Scholer SJ, Hudnut-Beumler J, Dietrich MS. The effect of physician--parent discussions and a brief intervention on caregivers' plan to discipline: is it time for a new approach? Clin Pediatr (Phila). 2011 Aug;50(8):712-9. doi: 10.1177/0009922811400730. Epub 2011 Mar 10. PMID 21393318
- [Background] Scholer SJ, Hudnut-Beumler J, Dietrich MS. A brief primary care intervention helps parents develop plans to discipline. Pediatrics. 2010 Feb;125(2):e242-9. doi: 10.1542/peds.2009-0874. Epub 2010 Jan 18. PMID 20083523
- See also: Access Play Nicely Multimedia Program — http://www.playnicely.org
- See also: AAP Connected Kids Program — http://www.aap.org/connectedkids/